CLINICAL TRIAL: NCT05206409
Title: Prediction of Delivery Mode by Ultrasound-assessed Fetal Position in Nulliparous Women With Prolonged First Stage of Labor.
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Other Study IDs: MS 747/2021
Record Dates: First submitted 2022-01-21; First posted 2022-01-25 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2022-01

CONDITIONS: Prolonged Labor
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Ultrasound — Fetal head position determination using ultrasound

SUMMARY:
In the past years, numerous studies have been published on the use of ultrasound during labor, showing this is an effective, accurate and objective tool for the assessment of the fetal head position and station. Literature affirmed that traditional transvaginal digital examination is highly subjective and dependent on the operator's experience. On the contrary, the use of intrapartum suprapubic transabdominal ultrasound can improve accuracy in determination of fetal head position and the precise knowledge of the location of specific fetal head landmarks in relationship to maternal pelvis. Intrapartum ultrasound will assist obstetricians in the diagnosis of normal labor progression, suggesting when medical and or operative intervention should be taken in case of complications.

ELIGIBILITY:
Inclusion Criteria:

* nulliparous women
* Singleton pregnancy
* prolonged first stage of Labor
* average fetal weight
* gestational age at or beyond 37 weeks

Exclusion Criteria:

* IUFD
* malpresentation

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Nulliparous women with delayed first stage of Labor
Sampling Method: Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2022-01-25 (Actual); Primary Completion 2023-08-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
Mode of delivery | 6 months
  Correlation between fetal head position and mode of delivery

CONTACTS AND LOCATIONS:
Locations (1):
- AinShams Maternity Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided